CLINICAL TRIAL: NCT05787613
Title: A Phase II Study to Evaluate the Efficacy, Safety and Tolerability of HLX26 (Anti-LAG-3 Monoclonal Antibody Injection) Combined With Serplulimab (Anti-PD-1 Humanized Monoclonal Antibody Injection) and Chemotherapy in Previously Untreated Advanced Non-small Cell Lung Cancer (NSCLC) Patients
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of HLX26 (Anti-LAG-3 Monoclonal Antibody Injection) Combined With Serplulimab and Chemotherapy in Previously Untreated Advanced NSCLC Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HLX26HLX10-NSCLC201
Record Dates: First submitted 2023-03-03; First posted 2023-03-28 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HLX26 MTD + serplulimab 300 mg + chemotherapy intravenous infusion Q3W (Experimental): In this group, HLX26 (MTD) in combination with HLX10 (300 mg) and chemotherapy will be intravenously administered every 3 weeks. About 40 subjects will be enrolled in this cohort. Patients will be treated with until disease progression, death, receiving new antitumor treatment, intolerable toxicity or withdrawal of informed consent (whichever occurs first). The efficacy of HLX26 (MTD) in combination with Serplulimab and chemotherapy will be evaluated in this group.
  Interventions: Drug: HLX26; Drug: Serplulimab; Drug: Chemotherapy drug
- HLX26 MTD-1 + serplulimab 300 mg + chemotherapy intravenous infusion Q3W (Experimental): In this group, HLX26 (MTD-1) in combination with HLX10 (300 mg) and chemotherapy will be intravenously administered every 3 weeks. About 40 subjects will be enrolled in this cohort. Patients will be treated with until disease progression, death, receiving new antitumor treatment, intolerable toxicity or withdrawal of informed consent (whichever occurs first). The efficacy of HLX26 (MTD-1) in combination with Serplulimab and chemotherapy will be evaluated in this group.
  Interventions: Drug: HLX26; Drug: Serplulimab; Drug: Chemotherapy drug
- placebo + serplulimab 300 mg + chemotherapy intravenous infusion Q3W (Placebo Comparator): In this group, placebo in combination with HLX10 (300 mg) and chemotherapy will be intravenously administered every 3 weeks. About 40 subjects will be enrolled in this cohort. Patients will be treated with until disease progression, death, receiving new antitumor treatment, intolerable toxicity or withdrawal of informed consent (whichever occurs first). The efficacy of Serplulimab and chemotherapy will be evaluated in this group.
  Interventions: Drug: Serplulimab; Drug: Chemotherapy drug; Drug: Placebo

INTERVENTIONS:
Drug: HLX26 — Anti-LAG-3 monoclonal Antibody Injection
  Other Names: Anti-LAG-3 monoclonal Antibody Injection
  Arms: HLX26 MTD + serplulimab 300 mg + chemotherapy intravenous infusion Q3W; HLX26 MTD-1 + serplulimab 300 mg + chemotherapy intravenous infusion Q3W
Drug: Serplulimab — anti-PD-1 humanized monoclonal antibody injection
  Other Names: HLX10
Drug: Chemotherapy drug — non-squamous NSCLC patients will receive Pemetrexed 500mg/m2, IV, Q3W. Carboplatin AUC 5mg/mL/min, IV, Q3W, up to 4 cycles.squamous NSCLC patients will receive Albumin-paclitaxel 100mg/m2, IV, Q1W or paclitaxel 175mg/m2, IV, Q3W and carboplatin AUC 5 mg/mL/min, IV, Q3W, up to 4 cycles.
Drug: Placebo — placebo
  Arms: placebo + serplulimab 300 mg + chemotherapy intravenous infusion Q3W

SUMMARY:
A Phase II Study to Evaluate the Efficacy, Safety and Tolerability of HLX26 (Anti-LAG-3 Monoclonal Antibody Injection) Combined With Serplulimab (Anti-PD-1 Humanized Monoclonal Antibody Injection) and Chemotherapy in Previously Untreated Advanced Non-small Cell Lung Cancer (NSCLC) Patients

DETAILED DESCRIPTION:
This study is a phase II study to evaluate the efficacy, safety and tolerability of HLX26 in combination with Serplulimab and chemotherapy in the treatment of patients with Non-small cell lung cancer.

The trial was divided into period 1 (safety run-in phase) and period 2 (dose expansion phase).

The first phase is an open-label study, patients will receive varying doses (800 mg, 600 mg or lower) of HLX26 combined with a fixed dose (300 mg) of serplulimab and chemotherapy, administered by intravenous infusion every 3 weeks. Observation period of DLT lasts for 3 weeks after the first administration of HLX26. Safety review committee (SRC) will responsible for the safety of combination treatment. After confirmation of the safety, the efficacy of HLX26 combined with Serplulimab and chemotherapy will be evaluated in period 2.

The second phase (dose expansion phase) is a randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of 2 dose levels of HLX26 combined with fixed-dose (300 mg) of serplulimab and chemotherapy in patients with NSCLC. If the tolerability observation of the 600mg dose group is completed in the first phase, the SRC will review the safety data obtained from the study and decide whether to enter into the second phase; if 2 of the 6 subjects in the 600mg dose group in the first phase occur DLT event, we will continue to explore the safe dose of HLX26 and enroll another 3-6 subjects. Once the maximum tolerated dose (MTD) is found, two doses, MTD and MTD-1, will be selected to enter the dose expansion phase. (The SRC will review the safety and tolerability results obtained in the study to determine the MTD, and will select the dose of MTD-1 below the MTD and within the effective dose range). In the second stage, there are 3 groups and 40 people in each group. The interactive network/voice response system (IWRS) is used to randomly assign qualified subjects to the following three groups in a 1:1:1 allocation ratio:

> Group A: HLX26 MTD intravenous infusion + serplulimab 300 mg intravenous infusion, Q3W; chemotherapy

> Group B: HLX26 MTD-1 intravenous infusion + serplulimab 300 mg intravenous infusion, Q3W; chemotherapy

> Group C: placebo + serplulimab 300 mg intravenous infusion, Q3W; chemotherapy

The chemotherapy will be decided by investigator per patients' pathological type. nsqNSCLC patients will receive pemetrexed and carboplatin as chemotherapy and sqNSCLC patients will receive nab-paclitaxel or paclitaxel and carboplatin.

ELIGIBILITY:
Key Inclusion Criteria:

1. Stage IV (AJCC 8th Edition) non-small cell lung cancer confirmed by histology or cytology.
2. No EGFR sensitive mutation or ALK, ROS1 rearrangement.
3. Have not received systemic treatment for stage IV disease. For patients who have received adjuvant or neoadjuvant treatment, if the adjuvant/neoadjuvant treatment has been completed for at least 6 months, they are allowed to be enrolled.
4. At least one measurable lesion evaluated by the investigator per RECIST v1.1.
5. Subjects must provide qualified tumor tissue samples for the detection of PD-L1 and LAG-3 expression level.
6. Have adequate organ function with expected survival period ≥ 12 weeks and ECOG score of 0 or 1.

Key Exclusion Criteria:

1. Subjects with other histopathological types including small cell lung cancer, neuroendocrine cancer or sarcoma.
2. Have other malignant tumors within 3 years.
3. Pleural effusion, pericardial effusion or ascites that require clinical intervention.
4. Myocardial infarction and poorly controlled arrhythmia occurred within six months before the first administration of the study drug.
5. III - IV cardiac insufficiency per NYHA standard or left ventricular ejection fraction<50%.
6. Patients with active pulmonary tuberculosis.
7. Patients with previous or current interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, or severe pulmonary function impairment that may interfere with the detection and management of suspected drug-related pulmonary toxicity.
8. Patients who have known active autoimmune diseases or suspected auto-immue disease. Patients in stable condition and do not require systemic immunosuppressant therapy are allowed to be enrolled.
9. Require systemic treatment with corticosteroids (> 10 mg/day prednisone or equivalent) or other immunosuppressive agents within 14 days prior to the first dose of the study products or during the study.
10. Patients who have received any T-cell costimulatory agents or immune checkpoint blockade therapy, including but not limited to cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) inhibitors, PD-1 inhibitors, PD-L1 inhibitors.
11. Patients with a history of severe allergy to any monoclonal antibody products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) (Part 1) | from day1 to day 21
  The DLT of HLX26 in combination with Serplulimab and Chemotherapy within 3 weeks after the first administration in previously untreated NSCLC patients
Maximum Tolerated Dose (MTD) (Part 1) | from day1 to day 21
  The MTD of HLX26 in combination with Serplulimab and Chemotherapy within 3 weeks after the first administration in previously untreated NSCLC patients
Objective Response Rate (ORR) per RECIST 1.1 as Assessed by IRRC ( Part 2) | approximately up to 12 months
  The ORR is defined as the percentage of participants who achieve a complete response (CR) or partial response (PR) per RECIST 1.1 as assessed by IRRC.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) per RECIST 1.1 assessed by IRRC and Investigator | approximately up to 12 months
Disease Control Rate (DCR) per RECIST 1.1 as Assessed by IRRC and Investigator | approximately up to 12 months
Duration of Response (DOR) per RECIST 1.1 assessed by IRRC and Investigator | approximately up to 12 months
Objective Response Rate (ORR) per RECIST 1.1 assessed by Investigator | approximately up to 12 months
  The ORR is defined as the percentage of participants who achieve a complete response (CR) or partial response (PR) per RECIST 1.1 as assessed by investigator.
Overall Survival (OS) | approximately up to 36 months
Adverse events | approximately up to 12 months
  The incidence of AE, SAE will be detected
Serum concentration of HLX26 and Serplulimab | approximately up to 12 months
  The serum concentration of HLX26 (at Cycle 1,2,4 and every 4 cycles from Cycle 8 and thereafter) and Serplulimab (at Cycle 4) will be detected.
Immunogenicity of HLX26 | approximately up to 12 months
  The incidence of Anti-HLX26 antibody and the incidence of neutralizing antibody will be detected

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No